CLINICAL TRIAL: NCT00957086
Title: Phase III, Double-Blind, Placebo-Controlled Study of Post-Operative Adjuvant Concurrent Chemo-Radiotherapy With or Without Nimotuzumab for Stage III/IV Head & Neck Squamous Cell Cancer
Brief Title: Study of Post-Op Adjuvant Concurrent Chemo-RT With or Without Nimotuzumab for Head & Neck Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IHN01
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Phase III Adjuvant Concurrent Chemo-RT +/- nimotuzumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab (Active Comparator): Comprising Adjuvant Cisplatin, Concurrent RT and Nimotuzumab
  Interventions: Drug: Nimotuzumab
- Placebo (Placebo Comparator): Comprising Adjuvant Cisplatin, Concurrent RT and Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — Administered by intravenous infusion at 200 mg absolute per dose, diluted in 250 ml of sodium chloride over 30 minutes. 8 weekly doses of study drug will be given, beginning on first week of radiotherapy.
  Arms: Nimotuzumab
Drug: Placebo — Administered by intravenous infusion at 200 mg absolute per dose, diluted in 250 ml of sodium chloride over 30 minutes. 8 weekly doses of study drug will be given, beginning on first week of radiotherapy.
  Arms: Placebo

SUMMARY:
The aim of the study is to improve the loco-regional control rate and overall survival of locally advanced head and neck squamous carcinoma (HNSCC). The investigators hypothesize that the addition of nimotuzumab (a recombinant humanized murine immune antibody that blocks both epidermal growth factor (EGF) and transforming growth factor (TGF)) to the current gold standard of concurrent chemoradiotherapy (CCRT) (7)(8), an adjuvant setting in patients after resection of their locally advanced HNSCC will confer therapeutic advantage.

DETAILED DESCRIPTION:
The aim of the study is to improve the loco-regional control rate and overall survival of locally advanced head and neck squamous carcinoma (HNSCC). We hypothesize that the addition of nimotuzumab (a recombinant humanized murine immune antibody that blocks both epidermal growth factor (EGF) and transforming growth factor (TGF)) to the current gold standard of concurrent chemoradiotherapy (CCRT) (7)(8), an adjuvant setting in patients after resection of their locally advanced HNSCC will confer therapeutic advantage. We have designed a phase III randomized study that includes a placebo arm. We assume a 10% increase in 2 year disease free survival (from 60% to 70%). To achieve statistical significance at 90% power, we calculate the need for 355 patients per arm, assuming also a 10% dropout rate. We aim to accomplish this study with the involvement of a multidisciplinary team of surgical, radiation and medical oncologists actively involved in the management of HNSCC coming from multiple institutions and spanning at least 12 different countries. For quality assurance we will have the involvement of Singapore Clinical Research Institute who will lead the data coordination and ensure fidelity of data collected and statistical analysis; the European Society of Therapeutic Radiation Oncology (EQUAL-ESTRO) for radiation dose and fields and an international independent panel of medical oncologist, radiation oncologist and biostatistician for the Data Monitoring Committee (DMC). This committee will monitor significant events and advise on continuation or termination of trial. Concurrent with the randomized trial, we will be collecting bio specimens including blood, tumour and saliva, pre-treatment and on completion of surgical resections. We hypothesize that there are important biomarkers including clusters of genes, cancer stem cells that will predict prognosis and treatment response. The analyses performed will be very powerful because of the large sample size, the specimens are collected prospectively and because the statistical analyses will be multivariate, incorporating not only treatment but biological and staging data.

ELIGIBILITY:
Inclusion Criteria:

* Age should be greater than or equal to the minimum age of consent in the applicable country
* Histologically proven head and neck squamous cell cancer (excluding nasopharynx, salivary glands, paranasal sinuses and unknown primaries) on biopsy of the primary lesion or the neck mass.
* Resectable stage III/IV according to the AJCC/UICC staging system with no evidence of distant metastasis.
* Complete macroscopic resection.
* Patients should have at least one of the following pathological features for inclusion: pT3 or pT4 and any nodal stage (N), except T3N0 of the larynx, with negative resection margins, or a tumor stage of 1 or 2 with a nodal stage of 2 or 3 and no distant metastasis (M0); patients with stage T1 or T2 and N0 or N1 who had unfavorable pathological findings (extranodal spread, positive resection margins, perineural involvement, or vascular tumor embolism) are also eligible, as are those with oral-cavity or oropharyngeal tumors with involved lymph nodes at level IV or V.
* Performance status must be ECOG 0 or 1. Patients should be able to tolerate chemotherapy and radiotherapy.
* Adequate bone marrow, renal and hepatic function:

  1. WBC>3000/mm3, platelets>100000/mm3
  2. Serum creatinine<upper limit of normal range as per institution and calculated creatinine clearance (according to the Cockcroft and Gault method) >50 ml/min.
  3. SAP, SGOT<2 x upper limit of normal range, bilirubin <1.5 x upper limit of normal range.
* Written informed consent.

Exclusion Criteria:

* Histology other than SCC or its subtype.
* Patients with disease subsite deemed suitable for organ preservation approach, namely stage III/IV laryngeal or hypopharyngeal carcinoma with not more than low-volume T4 disease; low-volume T4 disease is defined as disease not eroding into cartilage or extending not more than 1 cm into the base of tongue.
* Clinical or radiological evidence of distant metastasis.
* Uncontrolled comorbidities such as diabetes mellitis, hypertension, cardiac disease.
* Uncontrolled infection.
* Uncontrolled hypercalcemia.
* Prior history of cancer less than 5 years ago or a synchronous primary outside the head and neck area.
* Prior treatment, head and neck radiotherapy, chemotherapy or surgery (excluding biopsy) or anti-EGFR therapy such as cetuximab/EGFR oral tyrosine kinase inhibitor.
* Patients for whom compliance with follow-up is unlikely.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2009-08-13 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the disease-free survival between patients randomized to adjuvant nimotuzumab/cisplatin/RT with the control arm | 5 years

SECONDARY OUTCOMES:
To compare the overall survival between the two arms | 5 years
To assess the Toxicity Profile between the 2 arms | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: K C Soo, Prof, Study Chair — National Cancer Centre
Locations (30):
- Australia (2):
  - Flinders Medical Centre, Bedford Park
  - Peter MacCallum Cancer Centre, Melbourne
- National Institute of Oncology and Radiobiology, Vedado, Cuba
- Egypt (2):
  - Alexandria University School of Medicine, Alexandria
  - National Cancer Institute, Cairo University, Cairo
- India (6):
  - Apollo Hospital Bangalore, Bangalore
  - Narayana Hrudayalaya Hospital (Mazumdar Shaw Cancer Institute), Bangalore
  - Amrita Institute of Medical Sciences, Kerala
  - Tata Memorial Centre, Mumbai
  - Christian Medical College, Tamil Nadu
  - Regional Cancer Center Trivandrum, India, Trivandrum
- Cipto Mangunkusumo General Hospital Indonesia, Jakarta, Indonesia
- Malaysia (2):
  - Pantai Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Mahkota Medical Center, Malacca
- Philippines (2):
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
- King Fahad Medical City, Riyadh, Saudi Arabia
- National Cancer Centre, Singapore, Singapore
- South Africa (2):
  - The Oncology Centre, Durban
  - GVI Oncology, Panorama
- South Korea (4):
  - National Cancer Center Korea, Gyeonggi-do
  - INHA University Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taipei Med Univ Hosp [TMUH], Taipei
  - Taipei Veteran General Hospital, Taipei
- Thailand (3):
  - National Cancer Institute Bangkok (+Chulabhorn for RT), Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai Hospital, Chiang Mai